CLINICAL TRIAL: NCT04902547
Title: Evaluation of a Patient-Centred, Multidisciplinary Opioid Tapering Program for Individuals With Chronic Non-Cancer Pain on Long Term Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Dana Turcotte, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS23962
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use; Opioids; Harmful Use; Hyperalgesia; Pain, Chronic
Keywords: ACT; Opioid; Chronic Pain; Opioid Tapering; Opioid Stewardship; Pain Management
MeSH Terms: conditions — Hyperalgesia; Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either Multidisciplinary Tapering Program Only or Patient Education Workshops PLUS Multidisciplinary Tapering Program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Tapering Program Only (Experimental): Patients in this arm will take part in the clinical multidisciplinary opioid tapering program (MTP).
  Interventions: Procedure: Multidisciplinary Tapering Program
- Patient Education Workshop & Multidisciplinary Tapering Program (Experimental): As above, though patients in this group will also take part in an opioid education workshop
  Interventions: Behavioral: Patient Education Workshop (PEWs); Procedure: Multidisciplinary Tapering Program

INTERVENTIONS:
Behavioral: Patient Education Workshop (PEWs) — The comprehensive workshops will include a combination of didactic and interactive content on general pain and opioid education (1 hour workshop session to be co-presented by Drs Ryan Amadeo and Dana Turcotte) along with significant psychological content (co-presented by Drs Brigitte Sabourin and Gregg Tkachuk) making up the remainder of the day-long workshop. Content presented in PEWs will include opioid-related risks, identifying personal motivation for (or barriers to) tapering, goal setting, pain self-management, sleep hygiene and comprehensive focus on ACT and rethinking pain. During the interprofessionally co-facilitated sessions, participants will be provided with workbooks that will contain session specific content as well as take-home activities and information for their own personal use.
  Arms: Patient Education Workshop & Multidisciplinary Tapering Program
Procedure: Multidisciplinary Tapering Program — The MTP will begin with a Baseline Tapering Visit and will include the same baseline health and well-being questionnaires, a medication review, relevant pain history, relevant opioid use history, discussion re: patient-specific tapering and functional goals, taper start date, and determination if a different opioid formulation will be required for the taper. A detailed taper plan will be prepared and reviewed by the study clinician(s) and provided to the patient. In general, tapers will begin with a 10% reduction of dose every 2 weeks until ⅓ of the original dose is met, or until taper goal has been met. If further tapering is planned once the patient reaches ⅓ of their original dose, the taper will be reduced to half the volume and rate noted above in order to improve tapering success.
  Tapering plans and approaches may be changed (slowed, increased, halted etc.) based on follow up.

SUMMARY:
Chronic pain management is complex, with healthcare providers historically relying on prescribing opioid medications such as morphine. Although opioids may partially improve pain, there are risks associated with them as well, including pain worsening, side effects, addiction and overdose. It is now understood that the management of chronic pain is more effective when multiple healthcare team members work together and incorporate multiple strategies instead of focusing solely on medications. An example of an effective, non-drug strategy for pain is a service offered by clinical psychologists called "Acceptance and Commitment Therapy" - or ACT - which empowers individuals, to implement alternative ways of thinking about and reacting to pain and its effect on their lives.

Canada has responded to the opioid overdose crisis with new guidelines that encourage physicians and those suffering from chronic pain to aim for lower opioid doses whenever possible, a process often referred to as "tapering." Unsurprisingly, tapering opioids is often difficult for patients to consider, primarily due to misconceptions that it will cause more harm than good.

This project aims to address these misconceptions by developing and offering an all-day educational workshop for patients, co-presented by a healthcare team (clinical psychologists, pharmacists and physicians), to provide in-depth information on opioid related risks and misconceptions, as well as a large component focusing on ACT training. Investigators then want to see if these sessions change individual attitudes towards opioid tapering and if it improves willingness and ability to successfully reduce opioid doses to a safer level.

DETAILED DESCRIPTION:
Study Objectives:

1. To evaluate the impact of a patient-centered, multidisciplinary opioid tapering program on overall opioid consumption in individuals with chronic pain on long-term opioid therapy.
2. To implement opioid patient education workshops to be used in conjunction with the opioid tapering program and evaluate their preliminary feasibility and overall patient acceptance.

As Canada continues to witness a growing opioid crisis, the role of non-opioid medications and non-pharmacological strategies for pain, including behavioral treatments, is becoming more apparent. There is a great need to develop multidisciplinary clinical programs to assist individuals on long term opioid therapy to safely and effectively taper to safer doses of these potentially harmful medications. The use of nonpharmacological modalities will be integral to this process.

All patients enrolled in this project will be given the opportunity to take part in an informed and targeted multidisciplinary opioid tapering program (MTP). As well, half of the study population will be randomly assigned to also take part in a comprehensive opioid education and chronic pain workshop (Patient Education Workshop; PEW).

Abbreviated Methodology:

Individuals on LTOT at recruitment sites will be informed about the project by a member of their care team and those who show interest will be contacted and screened based on inclusion/exclusion criteria. Those who meet these criteria and consent to participate will be randomized to either the PEW + MTP cohort or the MTP only cohort. Depending on randomization, patients will then be invited to first attend a PEW or to attend a care visit to begin their tapering program. Participants completing the workshop will then begin the same tapering program at the MTP only cohort.

Multidisciplinary Tapering Program: Participants who have completed the Informed Consent Form ("MTP + PEW" and "MTP only" cohorts) will be included in the MTP, which will be conducted in collaboration with the patient's referring physician. All referring physicians from recruitment sites will be made aware of their role requirements in this study should their patients continue on to the MTP phase. Tapering programs will be individualized for all patients based on their current dose of opioid and clinical picture, and tapering planning will be co-managed by Drs. Amadeo and Turcotte, with the implementation and monitoring assistance of Pain Clinic nurses and Karin Ens (Clinical Pharmacist - ACCESS Winnipeg West). All participants will be asked to complete a battery of self-report measures of pain disability, pain, depression, anxiety, quality of life, pain acceptance, and valued living prior to the initiation of their tapering program (Baseline Visit) and again at 3-, 6-, and 12-month follow-up periods. Follow up has been identified as a crucial component of the MTP and will be managed by the clinical study team and clearly outlined in the detailed taper plan provided to referring physicians. Tapering plans and approaches may be changed (slowed, increased, halted etc.) based on results of this follow up at the discretion of study clinicians. Any changes/updates discussed with participants will be communicated to the referring physician with updated prescription or schedule changes. Like the tapering plan, the follow-up will be flexible and will depend on the patient's response to reductions and subsequent rate of taper. Follow up will include a combination of in-person and phone visits.

Patient Education Workshops: PEWs will be held as a full day session (approximately 9:30am to 3:30pm) and offerings will alternate between weekday and Saturday options to ensure flexibility for participants. Sessions will be offered monthly, or more often if the demand exists. The PEWs have been developed through a highly collaborative and interprofessional process and include some adaptations of previous work (used with permission) in order to create a session that is multidisciplinary, patient-centred and applicable to various forms of CNCP. The comprehensive workshops will include a combination of didactic and interactive content on general pain and opioid education (1 hour workshop session to be co-presented by Drs Ryan Amadeo and Dana Turcotte, and Karin Ens) along with significant psychological content (co-presented by Drs Brigitte Sabourin and Gregg Tkachuk) making up the remainder of the day-long workshop. Content presented in PEWs will include opioid-related risks, identifying motivation for (or barriers to) tapering, goal setting, pain self-management, sleep hygiene and comprehensive focus on ACT and rethinking pain. During the interprofessionally co-facilitated sessions, participants will be provided with workbooks that will contain session specific content as well as take-home activities and information for their own use.

Study Significance: The project will develop educational material aimed at furthering the understanding of both appropriate and inappropriate opioid prescribing in CNCP. This material will be available for consumption, beyond the project, with the knowledge users described. This will be undertaken at academic conferences, as well as at administrative gatherings in both academic and clinical settings. The knowledge created from this project, both in the program undertaken as well as in the collection and analysis of the endpoints outline, will allow for improved dialogue at all levels of health care. Both in the care of individual patients and in the public health approach to LTOT and opioid weaning, there will be improved understanding and process that will be accessible in broader primary care environments.

ELIGIBILITY:
Inclusion Criteria:

* CNCP on more than half the days in the previous 6 months
* use of opioids for more than half the days in the previous 90 days
* daily morphine equivalent dose equal to or greater than 50 mg
* age 18 years or older
* cognitive ability to understand questionnaires and participate in English only education sessions
* minimum average numerical pain rating of 3/10

Exclusion Criteria:

* Currently receiving ACT or CBT
* previous experience with ACT within the past 12 months
* significant uncontrolled depression with or without suicidal ideation
* current psychosis
* known or suspected opioid misuse/abuse based on a score of seven or greater on the Opioid Risk Tool
* known or suspected opioid diversion based on previous clinician report and/or results of urine drug screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Opioid use | Longitudinally, occurring at weekly/biweekly phone check-ins & in person visits at 0,3,6 and 12 months
  Using morphine equivalent doses, changes in opioid use will be evaluated
Pain level | Longitudinally, occurring at weekly/biweekly phone check-ins & in person visits at 0,3,6 and 12 months
  Using VAS tool, changes in pain will be evaluated

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - ACCESS River East, Winnipeg, Manitoba
  - ACCESS Winnipeg West, Winnipeg, Manitoba
  - Health Sciences Centre Pain Clinic, Winnipeg, Manitoba
  - Pan Am Pain Clinic, Winnipeg, Manitoba